CLINICAL TRIAL: NCT04982497
Title: Development and Evaluation of a Psychological Intervention in Videogame Format for the Promotion of Active Aging
Acronym: GAMEPROAGING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: State Research Agency, Spain (Other Government)
Responsible Party: Principal Investigator, Fernando Lino Vázquez González, Full Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PID2019-105052RB-I00
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Aging; Aging Problems
Keywords: video game; older adults; active aging; health promotion; study protocol
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video game based intervention (Experimental): The participants in the experimental group will receive a cognitive-behavioral intervention for active aging via an interactive online multimedia video game with a complementary App. The intervention will consist of 8 modules each approximately 70 (±25) minutes long that will be administered at a rate of 1 per week with between-session homework.
  Interventions: Behavioral: Video game based intervention
- Control group (Active Comparator): Individuals assigned to this group will receive online therapeutically inactive information about active aging.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Video game based intervention — The intervention will be administered via an online graphic-adventure video game. It includes 3 components: depression prevention, cognitive stimulation, and healthy habits promotion. The depression prevention component will be adapted from an indicated prevention program based on the model by Lewinsohn et al. (1985). The cognitive stimulation component is based on cognitive reserve (Tucker & Stern, 2011) and neuroplasticity (Shapiro, 2001), the cognitive stimulation model by Spector et al. (2006), and the causes of age-related memory failures (Light, 1991) (e.g., decrease in the processing resources, semantic coding deficit, difficulties in deliberate information retrieval). The healthy habits promotion component is based on the social learning and social cognitive theories (Bandura, 1986; Spiegler, 2016).
  Arms: Video game based intervention
Other: Control group — The active control group will have access to a platform of online therapeutically inactive information related to active aging.
  Arms: Control group

SUMMARY:
The social and health challenges of the aging population have led to the recommendation of active aging programs to increase the number of healthy and independent elderly people. These interventions have been shown to offer benefits in terms of quality of life, wellbeing, dietary and physical exercise habits, and cultural and social activity. However, there is a current need to investigate more-effective alternative means to disseminate these interventions beyond in-person formats such as serious videogames, aimed at promoting behavioral changes and providing education for purposes such as health or learning. The main objective of this project is to improve on a videogame intervention for the promotion of aging and to evaluate its efficacy via a randomized controlled trial. It is expected that after the intervention and in the follow-ups (at 3, 6, and 12 months), participants in the videogame arm of the study will have higher health status compared to the control group subjects. The first months of the study will be devoted to revising the materials and fine-tuning the intervention tested in a previous pilot study. After that, the randomized controlled trial will be conducted. Participants will be recruited through clinics and health care centers in the Autonomous Community of Galicia (Spain). To participate in the study, participants must: (a) be at least 45 years old, (b) have normal cognitive functioning, and (c) reside in Galicia. Participants will be excluded if they: (a) have serious mental or medical disorders; (b) have been receiving psychological or psychopharmacological treatment during the two months prior to the study or are participating in other studies related to active aging; and finally, (c) do not have the appropriate devices to play the game, cannot communicate in Spanish, or have problems that make it impossible to play the videogame. Information on various sociodemographic and clinical variables will be collected during the pre-intervention evaluation. The main outcome will be perceived health status, as evaluated using the SF-36 health questionnaire. A total of 548 participants will be randomly assigned to a cognitive-behavioral intervention administered through a serious online interactive multimedia game with a complementary App (CBI-V, experimental group) or to a control group that will receive information on active aging in an online format (CG). The randomization sequence will be generated automatically by the evaluation platform (concealment or blinding of randomization), and the participants in the CBI-V group will be given access to the first module of the intervention, while those in the CG will receive the first informational module. The participants in both groups will then complete the next seven modules for each condition. After the intervention, the participants will be evaluated in the postintervention assessment and follow-up assessments at 3, 6 and 12 months. In terms of its impact, this study will contribute to the development and rigorous evaluation of the worlds first psychological intervention to promote active aging managed through an interactive online multimedia videogame with a complementary app. In addition, confirmation of the programs clinical validity will be of great relevance in terms of health, social and economic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 45 years old.
* Have normal cognitive functioning.
* Reside in the region of Galicia (Spain).

Exclusion Criteria:

* Have serious mental or medical disorders (e.g., severe depression, schizophrenia, bipolar disorder, dementia, dissociative disorders, substance dependence, acute suicidal ideation).
* Recent psychological or psychiatric treatment (in the past 2 months), or participation in another trial related to active aging.
* Do not have the appropriate devices to play the game (computer and smartphone with internet connection), cannot communicate in Spanish, or have problems (e.g., sensory, physical) that make it impossible to play the videogame.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Health Status to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  Health status will be measured with the 36-Item Short-Form Health Survey [SF-36] (SF-36; Ware & Shebourne, 1992; Spanish version by Alonso et al., 1995 ). This is a self-administered measure that assesses perceived health status. It contains 36 items that form 8 dimensions: General health, Physical functioning, Physical role functioning, Bodily pain, Vitality, Social functioning, Emotional role functioning, and Mental health. The 8 dimensions are obtained by recalibrating scores for 10 items, computing raw scales, and transforming them to a 0-100 scale. Dimension scores range from 0 to 100, with higher scores indicating better health status. Their internal consistencies (Cronbach's alphas) range from .71 to .94. These dimensions can be combined in two factors (Physical health and Mental health) with an average of 50 and a standard deviation of 10, and internal consistencies of .94 and .89, respectively.

SECONDARY OUTCOMES:
Change from baseline Emotional distress to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  This will be measured with the General Health Questionnaire (GHQ-12; Goldberg & Williams,1988; Spanish version by Rocha et al., 2011). This self-administered questionnaire consists of 12 items and assesses emotional distress. The person evaluates each item based on their emotional distress using a Likert scale with four response options ranging from "better than usual" to "much worse than usual," which are scored using a bimodal response scale (0, 0, 1, 1). The total score ranges from 0 to 12, with higher scores indicating greater emotional distress. The internal consistency (Cronbach's alpha) is .86 for people under 65 and .90 for people 65 and older.
Change from baseline Depressive symptomatology to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  Depressive symptoms as measured by the Center for Epidemiological Studies Depression Scale (CES-D; Radloff, 1977; Spanish version by Vázquez et al., 2007). This 20- item scale is self-administered and assesses depressive symptoms. The person evaluates each item based on how often they have experienced it in the last week using a Likert scale with four response options ranging from 0 (rarely or none of the time) to 3 (most of the time). The total score ranges from 0 to 60, where higher scores correspond to greater depressive symptomatology. Internal consistency (Cronbach's alpha) of the scale is .89.
Change from baseline Reinforcement to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  To evaluate the reinforcement, we will use the Environmental Reward Observation Scale (EROS; Armento & Hopko, 2007; Spanish version by Barraca & Pérez-Álvarez, 2010). It is a self-administered 10-item scale that assesses the degree of positive reinforcement contingent on the response received from the media. Each item is evaluated based on the degree to which the individual believes applies to them, according to a Likert scale with four response options ranging from 1 (strongly disagree) to 4 (strongly agree). The total score ranges from 10 to 40, with higher scores indicating more positive reinforcement. The internal consistency (Cronbach's alpha) of the Spanish version is .86.
Change from baseline Negative automatic thoughts to post-treatment (9 weeks), and follow- ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  The occurrence of automatic negative thoughts will be assessed through the Automatic Thoughts Questionnaire (ATQ; Hollon & Kendall, 1980; Spanish version by Otero et al., 2017). This is a 30-item self-report questionnaire that assesses negative thoughts. The subject must indicate the frequency for which a number of thoughts have suddenly arisen in their mind over the last week on a five-point scale from 1 (never) to 5 (always). Scores range between 30 and 150, with a higher score indicating more negative thoughts experienced by the subject. The ATQ's internal consistency (Cronbach's alpha) is .96.
Change from baseline Self-reported memory to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  Self-reported memory will be measured with the Multifactorial Memory Questionnaire (MMQ; Troyer & Rich, 2002). This 57-item self-administered test assesses subjective memory. Items are rated on a 5-point Likert scale based on the test taker's experiences over the previous two weeks. It comprises three dimensions: Contentment, Ability, and Strategy. Contentment measures satisfaction, concern, and overall appraisal of one's own memory; the score ranges from 0 to 72, with higher scores indicating greater satisfaction. The internal consistency is .95. Ability measures self-perception of everyday memory ability; the score range is 0 to 80, with higher scores indicating better self-reported memory ability, with an internal consistency of .93. Strategy measures the use of practical memory strategies in day-to-day life; the score range is 0 to 76, with higher scores indicating greater use of memory strategies. The internal consistency is .83.
Change from baseline Sleep hygiene behaviors to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  Participants' sleep hygiene behaviors will be assessed with the Sleep Hygiene Index (SHI; Mastin et al., 2006). It is a 13-item self-report measure designed to assess the practice of sleep hygiene behaviors. Each item is rated on a five-point scale ranging from 0 (never) to 4 (always). The total score ranges from 0 to 52, with a higher score representing poorer sleep hygiene. Its internal consistency (Cronbach's alpha) is .66.
Change from baseline Physical Activity to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  Participants' physical activity will be assessed with the Brief Physical Activity Assessment Tool (BPAAT; Marshall et al., 2005; Spanish version by Puig et al., 2012). This two-item questionnaire measures the frequency and duration of moderate and vigorous physical activity in an individual's usual week. Combining the results of both questions, scores can range from 0 to 8, with a higher score indicating higher physical activity. In addition, the subject can be classified as sufficiently (≥4 score) or insufficiently active (0-3 score). The questionnaire has good test-retest reliability and content validity.
Change from baseline Eating habits to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  Eating habits will be assessed with the Rapid Eating and Activity Assessment for Participants-Shortened Version (REAP-S; Segal-Isaacson et al., 2004 ). This 16-item scale assesses the consumption of different food groups. The total score ranges from 13 to 39, with a higher score representing better eating habits. This instrument has shown good convergent validity with the Block Semi Quantitative Food Frequency Questionnaire (Block, 1998), and is based on the Dietary Guidelines of the U.S. Department of Health and Human Services (Office of Disease Prevention and Health Promotion, 2015 ) and the Healthy People 2010 objectives (U.S.Department of Health and Human Services, 2000 ).
Change from baseline Body Mass Index to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  The Body Mass Index (BMI) is a measure of nutritional status in adults. It is defined as an individual's weight in kilograms divided by the square of the height in meters (kg/m2) and classifies nutritional status as underweight, normal weight, pre-obesity, and obesity (I, II, and III).
Change from baseline Social support to post-treatment (9 weeks), and follow-ups at 3, 6 and 12 months | Pre- and post-intervention (9 weeks) with follow-ups at 3, 6 and 12 months
  Social support will be assessed with the Duke-UNC Functional Social Support Questionnaire (Duke-UNC-11; Broadhead et al., 1988 ; Spanish version by Bellón et al., 1996). This self-report 11-item test assesses perceived social support. Each item is rated on a 5-point scale ranging from 1 (never) to 5 (always). The total score ranges from 11 to 55, with a higher score representing more social support. Its internal consistency (Cronbach's alpha) is .90.
Dropouts and treatment adherence | During the intervention sessions (8 weeks)
  Dropouts will be assessed by means of a register throughout the study. Treatment adherence will be automatically registered using both the online video game and the App by means of the number of modules completed by each participant, the time played, the time spent on cognitive tasks throughout the game and between session homework accomplishment.
Satisfaction with the service received | Post-intervention (9 weeks)
  Participant satisfaction with the service received will be evaluated upon intervention completion. We will use the Client Satisfaction Questionnaire (CSQ-8; Larsen et al., 1979; Spanish version by Vázquez et al., 2017). It is a 8-item scale with 4 possible answers and a final ranking score ranging from 8 to 32, where a higher score implies greater satisfaction with the service received. It has an internal consistency of .80.

OTHER OUTCOMES:
Socio-demographic characteristics | Pre-intervention
  Sociodemographic characteristics will be collected through a questionnaire elaborated ad hoc for this study. Participant data will include sex, age, marital status, level of education, main occupation and family monthly income per household.
Cognitive function | Screening
  Cognitive function will be assessed with the Mini-mental State Examination (MMSE; Folstein et al., 1975; Spanish version by Lobo et al., 1999). This 30-item instrument is used extensively in clinical and research settings to measure cognitive impairment. It has norms adjusted for age and education, good reliability values, and a sensitivity of 89.8% and specificity of 75.1%.
Diagnostic Interview | Screening
  For the diagnostic interview, the Mini International Neuropsychiatric Interview (M.I.N.I.; Sheehan et al., 1998; Spanish version by Ferrando et al., 2000) will be used. This diagnostic interview with 120 items explores the main mental disorders of Axis I of the Diagnostic and Statistical Manual (DSM-IV) or International Classification Diseases (ICD-10) and must be applied by a clinician. It has adequate reliability (k = 0.50-0.90), a sensitivity between 17%-92% and specificity of 75%-100%.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L. Vázquez González, PhD., Principal Investigator — University of Santiago de Compostela; Ángela J. Torres Iglesias, PhD., Principal Investigator — University of Santiago de Compostela
Locations (1):
- Research Group on Mental Health and Psychopatology, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
Researchers will report study results through publications. The data supporting these findings will be presented in the main publications, and the datasets used during the study can be obtained from the corresponding author on reasonable request.

REFERENCES:
- [Background] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470
- [Background] Armento ME, Hopko DR. The Environmental Reward Observation Scale (EROS): development, validity, and reliability. Behav Ther. 2007 Jun;38(2):107-19. doi: 10.1016/j.beth.2006.05.003. Epub 2006 Dec 12. PMID 17499078
- [Background] Bandura A. Social foundations of thought and action: A social cognitive theory: Englewood Cliffs, NJ, US: Prentice-Hall, Inc; 1986.
- [Background] Barraca J, Pérez-Álvarez M. Adaptación española del Environmental Reward Observation Scale (EROS) [Spanish adaptation of the Environmental Reward Observation Scale (EROS)]. Ansiedad Estrés 16:95-107, 2010.
- [Background] Bellon Saameno JA, Delgado Sanchez A, Luna del Castillo JD, Lardelli Claret P. [Validity and reliability of the Duke-UNC-11 questionnaire of functional social support]. Aten Primaria. 1996 Sep 15;18(4):153-6, 158-63. Spanish. PMID 8962994
- [Background] Block G. Invited commentary: comparison of the Block and the Willett food frequency questionnaires. Am J Epidemiol. 1998 Dec 15;148(12):1160-1; discussion 1162-5. doi: 10.1093/oxfordjournals.aje.a009601. No abstract available. PMID 9867260
- [Background] Broadhead WE, Gehlbach SH, de Gruy FV, Kaplan BH. The Duke-UNC Functional Social Support Questionnaire. Measurement of social support in family medicine patients. Med Care. 1988 Jul;26(7):709-23. doi: 10.1097/00005650-198807000-00006. PMID 3393031
- [Background] Ferrando L, Bobes J, Gibert J, Soto M, Soto O. MINI. Entrevista Neuropsiquiátrica Internacional. Versión en Español 5.0. [MINI. International Neuropsychiatric Interview. Spanish version 5.0] Madrid: Instituto IAP; 2000.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Goldberg D, Williams P. A user's guide to the General Health questionnaire. Windsor, UK: NFER-Nelson. 1988.
- [Background] Hollon SD, Kendall PC. Cognitive self-statements in depression: development of an Automatic Thoughts Questionnaire. Cognit Ther Res 4:383-95, 1980.
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Lewinsohn PM, Hoberman H, Teri L, Hautzinger M. An integrative theory of depression. In: Reiss S, Bootzin RR, editors. Theoretical issues in behaviour therapy. New York: Academic Press; 1985. p. 331-59.
- [Background] Light LL. Memory and aging: four hypotheses in search of data. Annu Rev Psychol. 1991;42:333-76. doi: 10.1146/annurev.ps.42.020191.002001. No abstract available. PMID 2018397
- [Background] Lobo A, Saz P, Marcos G, Dia JL, de la Camara C, Ventura T, Morales Asin F, Fernando Pascual L, Montanes JA, Aznar S. [Revalidation and standardization of the cognition mini-exam (first Spanish version of the Mini-Mental Status Examination) in the general geriatric population]. Med Clin (Barc). 1999 Jun 5;112(20):767-74. Spanish. PMID 10422057
- [Background] Marshall AL, Smith BJ, Bauman AE, Kaur S. Reliability and validity of a brief physical activity assessment for use by family doctors. Br J Sports Med. 2005 May;39(5):294-7; discussion 294-7. doi: 10.1136/bjsm.2004.013771. PMID 15849294
- [Background] Mastin DF, Bryson J, Corwyn R. Assessment of sleep hygiene using the Sleep Hygiene Index. J Behav Med. 2006 Jun;29(3):223-7. doi: 10.1007/s10865-006-9047-6. Epub 2006 Mar 24. PMID 16557353
- [Background] Office of Disease Prevention and Health Promotion. Dietary guidelines for Americans. Available from: http://www.health.gov/dietaryguidelines. [Accessed on 7th July 2021]
- [Background] Otero P, Vázquez FL, Blanco V, Torres A. Propiedades psicométricas del Cuestionario de Pensamientos Automáticos (ATQ) en cuidadores familiares [Psychometric properties of the Automatic Thoughts Questionnaire (ATQ) in family caregivers]. Behav Psychol. 25, 387-403, 2017.
- [Background] Puig Ribera A, Pena Chimenis O, Romaguera Bosch M, Duran Bellido E, Heras Tebar A, Sola Gonfaus M, Sarmiento Cruz M, Cid Cantarero A. [How to identify physical inactivity in primary care: validation of the Catalan and Spanish versions of 2 short questionnaires]. Aten Primaria. 2012 Aug;44(8):485-93. doi: 10.1016/j.aprim.2012.01.005. Epub 2012 Mar 29. Spanish. PMID 22463945
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement. 1977; 1:385-401
- [Background] Rocha KB, Pérez K, Rodríguez-Sanz M, Borrell C, Obiols JE. Propiedades psicométricas y valores normativos del General Health Questionnaire (GHQ-12) en población general española [Psychometric properties and normative values of the General Health Quationnnaire (GHQ-12) for Spanish population]. International Journal of Clinical and Health Psychology. 11(1), 125-139, 2011.
- [Background] Segal-Isaacson CJ, Wylie-Rosett J, Gans KM. Validation of a short dietary assessment questionnaire: the Rapid Eating and Activity Assessment for Participants short version (REAP-S). Diabetes Educ. 2004 Sep-Oct;30(5):774, 776, 778 passim. doi: 10.1177/014572170403000512. No abstract available. PMID 15510530
- [Background] Shapiro M. Plasticity, hippocampal place cells, and cognitive maps. Arch Neurol. 2001 Jun;58(6):874-81. doi: 10.1001/archneur.58.6.874. PMID 11405801
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Spector A, Thorgrimsen L, Woods RT, Orrell M. Making a difference: an evidence-based group programme to offer Cognitive Stimulation therapy (CST) to people with dementia. London, UK: Hawker Publications. 2006.
- [Background] Spiegler MD. Contemporary behavior therapy. Boston, US: Cengage Learning. 2016.
- [Background] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Background] Tucker AM, Stern Y. Cognitive reserve in aging. Curr Alzheimer Res. 2011 Jun;8(4):354-60. doi: 10.2174/156720511795745320. PMID 21222591
- [Background] US Department of Health and Human Services: Healthy People 2010. https://www.cdc.gov/nchs/healthy_people/hp2010/hp2010_final_review.htm. 2000. [Accessed on 7th July 2021]
- [Background] Vazquez FL, Blanco V, Lopez M. An adaptation of the Center for Epidemiologic Studies Depression Scale for use in non-psychiatric Spanish populations. Psychiatry Res. 2007 Jan 15;149(1-3):247-52. doi: 10.1016/j.psychres.2006.03.004. Epub 2006 Dec 1. PMID 17141880
- [Background] Vázquez FL, Torres Á, Otero P, Blanco V, Attkisson CC. Psychometric Properties of the Castilian Spanish Version of the Client Satisfaction Questionnaire (CSQ-8). Current Psychology 1(1): 1-7, 2017.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914